CLINICAL TRIAL: NCT02003313
Title: Immunogenicity and Safety of Group A, C, Y and W135 Meningococcal Polysaccharide Vaccine in More Than 2 Years Old Children and Adults
Brief Title: Immunogenicity and Safety of Group A, C, Y and W135 Meningococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012L02647; 2012L02647 (Registry Identifier: China food and drug administration)
Record Dates: First submitted 2013-11-28; First posted 2013-12-06 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Meningitis
Keywords: safety, immunogenicity, Meningococcal Polysaccharide Vaccine
MeSH Terms: conditions — Meningitis | interventions — Sensitivity Training Groups; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group T (Experimental): Participants of enrollment will receive 1 dose on Group A, C, Y and W135 Meningococcal Polysaccharide Vaccine.
  Interventions: Biological: Group T
- Group C (Active Comparator): Participants of enrollment will receive 1 dose on Group A, C, Y and W135 Meningococcal Polysaccharide Vaccine.
  Interventions: Biological: Group C

INTERVENTIONS:
Biological: Group T — 0.5ml, Intramuscular
  Other Names: vaccine made by Beijing Minhai Biotechnology Co., Ltd
  Arms: Group T
Biological: Group C — 0.5ml, Intramuscular
  Other Names: vaccine made by Hualan Biological Engineering, INC
  Arms: Group C

SUMMARY:
The purpose of this double-blind study is to evaluate the safety, reactogenicity and immunogenicity of Group A,C,Y and W135 Meningococcal Polysaccharide Vaccine in 2 to 30 years-old Children and Adults. All subjects will receive 1 dose of Group A,C,Y and W135 Meningococcal Polysaccharide Vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol should be enrolled in the study.
* Healthy permanent residence 2-30 years old.
* Subjects and parent/guardian able to attend all scheduled visits and comply with all study procedures.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* History of meningitis infection or vaccination of meningococcal vaccine within the past 6 months.
* Allergic history or any SAE after vaccination, such as allergy, urticaria, dyspnea, angioedema, celialgia.
* Patients administered with immunosuppressive agents, cytotoxicity factor or corticosteroids in the 6 months preceding the vaccine trial.
* Receipt of blood or blood-derived products in the 3 months preceding vaccination.
* Participation in another clinical study investigating a vaccine, drug in the 30 days preceding vaccination.
* Receipt of any live virus vaccine in the 15 days preceding vaccination.
* Receipt of any subunit vaccine and inactivated vaccine in the 7 days before vaccination.
* Febrile illness (temperature ≥ 38°C) in the 3 days or any acute illness/infection in the 7 days preceding vaccination.
* Thrombocytopenia.
* History of thyroid gland excision or treatment for thyroid gland disease in last 12 months.
* Functional or anatomic asplenia.
* History of eclampsia, epilepsy, encephalopathy and mental disease or family disease.
* Chronic disease (such as Down syndrome, diabetes, sickle cell anemia or neurologic disease, Guillain-Barre Syndrome).
* Known or suspected diseases, including: respiratory system disease, acute infection or active stage of chronic disease, HIV infection of children or mothers, cardiovascular disease, acute hypertension, cancer treatment, skin disease, etc.
* In pregnancy or lactation or pregnant women during the test plan
* Any condition that, in the judgment of investigator, may affect trial assessment.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1260 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects exhibiting a >=4 fold increase in rSBA titers level from pre-vaccination to post-vaccination | 28 days after vaccination

SECONDARY OUTCOMES:
to evaluate the adverse reactions after vaccination | within 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: nianmin shi, Principal Investigator — Beijing chaoyang district center for disease control and prevention
Locations (1):
- Chaoyang District Centre for Disease Prevention and Control, Beijing, China